CLINICAL TRIAL: NCT05603364
Title: Effect of Postoperative Oral Carbohydrate Administration in Total Knee Arthroplasty Elderly Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nanjing First Hospital Han Liu
Record Dates: First submitted 2022-10-16; First posted 2022-11-02 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2022-10

CONDITIONS: Total Knee Arthroplasty; Postoperative Oral Carbohydrates; Postoperative Recovery; Elderly Patients
MeSH Terms: interventions — maltodextrin; Fructose; Glucose

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EOF group：early carbohydrate feeding (Experimental): The EOF group drank 10.5% of 5 ml/kg body weight (100ml containing 12.5g maltodextrin, fructose and glucose) after extubation in the resuscitation room.
  Interventions: Combination Product: 100ml carbohydrate containing 12.5g maltodextrin, fructose and glucose
- Control group：conventional feeding (Experimental): Patients in group C were observed with 60minutes of abnormal vital signs after extubation, and returned to the ward for fasting and fasting for at least 6 hours, and began to eat gradually through the mouth after anal exhaust.
  Interventions: Other: Routine feeding

INTERVENTIONS:
Combination Product: 100ml carbohydrate containing 12.5g maltodextrin, fructose and glucose — Drank 10.5% of 5 ml/kg body weight (100ml containing 12.5g maltodextrin, fructose and glucose) after extubation in the resuscitation room.
  Arms: EOF group：early carbohydrate feeding
Other: Routine feeding — Patients in group C were observed with 60min of abnormal vital signs after extubation, and returned to the ward for fasting and fasting for at least 6 h, and began to eat gradually through the mouth after anal exhaust
  Arms: Control group：conventional feeding

SUMMARY:
To evaluate the effects of early oral carbohydrates after TKA on nutritional status, comfort and safety in elderly patients.

DETAILED DESCRIPTION:
Most of the current clinical studies of oral carbohydrate effects on postoperative recovery focus on the preoperative oral phase, and only a few small samples have shown that postoperative oral carbohydrate improves postoperative comfort. Therefore, further systematic studies on the effects of early postoperative oral carbohydrates on postoperative recovery remain lacking.

This clinical study uses a single center, randomized, single-blind, parallel controlled trial design divided into screening, treatment and follow-up period.

Actively control blood pressure, blood pressure and blood sugar, correct anemia and hypoproteinemia, and increase protein intake before surgery. The dietary plan was informed by the ward nurse: all patients were fasted with solid food 6 hours before surgery and took 200 milliliters of carbohydrates orally 2-3 hours before surgery.

The venous access was open after home invasion and was routinely monitored electrocardiogram (ECG), non-invasive blood pressure (NBP) ，oxygen saturation (SpO2) ，bispectral index (BIS). Parecoxib 40 milligrams of analgesia was given intravenously at 30 minutes before the start of the procedure. Adductor canal block (ACB) and Infiltration between popliteal artery and capsule of knee (IPACK) block were performed on the lower limbs of the surgical side using an ultrasound high-frequency line array probe before induction of the general anesthesia procedure.

Anesthesia induction: after static injection of Midazolam 0.03 milligrams / kilogram, Propofol 2 milligrams / kilogram， Sufentanyl 0.4 milligrams / kilogram, Cisatracurium 0.2 milligrams / kilogram. The tracheal tube was inserted after 3minutes and mechanical controlled ventilation was performed mechanical controlled ventilation, fraction of inspired oxygen（FiO2） 40%, oxygen flow 2 liters/ minutes, minute ventilation 7 milliliters / kilogram, respiratory rate（RR）12 times/ inspiration-to-expiratory ratio（I: E）1:2, maintain partial pressure of carbon dioxide in end expiratory gas （PETCO2） 35-40 millimeters of mercury（mmHg）. Anesthesia maintenance: intravenous propofol 4~7 milligrams / kilogram/ hour, remifentanil 0.3-0.5micrograms /kilogram/ hour, maintain BIS 40~60. A restrictive fluid management strategy was adopted, with 6ml/ kg·h supplemented with physiological needs, blood loss was supplemented with hydroxyethyl starch fluid, and concentrated red blood cells were infused at hemoglobin (Hb) <80 grams / litre to maintain patient blood pressure and heart rate fluctuations less than ±20% of the basal value. Dexamethasone 5mg and Tropisetron 2mg for prophylactic antiemesis were given intravenously at 30min before the end of the surgery. All patients used hydromorphone patient-controlled intravenous analgesia（PCIA ） pump for continuous: 1ml / h, automatic control: 5ml, locking: 10min, limit: 35ml / h, adjust parameters according to the pain.

Internal post anesthesia care unit （PACU） management: Patients will randomly enter the PACU into two study groups: early carbohydrate feeding group (EOF group) and conventional feeding group (control group). Routine feeding group (Group C): Patients in group C were observed with 60min of abnormal vital signs after extubation, and returned to the ward for fasting and fasting for at least 6 h, and began to eat gradually through the mouth after anal exhaust. Early carbohydrate feeding group (EOF group): The EOF group drank 10.5% of 5 ml/kg body weight (100ml containing 12.5g maltodextrin, fructose and glucose) after extubation in the resuscitation room. PACU management: Patients will randomly enter the PACU into two study groups: early carbohydrate feeding group (EOF group) and conventional feeding group (control group). Routine feeding group (Group C): Patients in group C were observed with 60min of abnormal vital signs after extubation, and returned to the ward for fasting and fasting for at least 6 h, and began to eat gradually through the mouth after anal exhaust. Early carbohydrate feeding group (EOF group): The EOF group drank 10.5% of 5 ml/kg body weight (100ml containing 12.5g maltodextrin, fructose and glucose) after extubation in the resuscitation room.

To evaluate the drinking criteria for patients in the EOF group: Steward wake score of 6 and wake level 3, take 5 ml/kg body weight of 12.5% carbohydrate (100ml containing 12.5g maltodextrin, fructose, and glucose) according to the patient's consent. The process of drinking carbohydrates was to take 30ml orally first. After observing the swallowing without abnormality, the patient was ordered to drink the remaining drinks within 2h. After the patient returns to the ward, the liquid diet is gradually excessive to the normal diet. When the patient was able to tolerate the normal diet, v.

1. Steward score: Awakening degree: 0-no response to stimulus; 1-some response to stimulus; 2-full awake.(2) Respiratory tract patency degree: 0 points-the patient's respiratory tract needs support; 1 points-the patient's respiratory tract can maintain patency without support; 2 points-the patient can cough according to the doctor's guidance.(3) Body activity degree: 1 points-the patient's limb has no activity; 2 points-the patient's limb has an unconscious activity; 3 points-the patient's limb can carry out conscious activities
2. Wakefulness classification according to the patient's consciousness performance: Level 0: the patient is completely asleep, Call without any response; Level 1: The patient is falling asleep, However, head and neck movement, eye opening or limb movement when breathing; level 2: the patient is awake, Have the same performance as level 1, At the same time can also open the mouth, stretch the tongue; Level 3: The patient is awake, Have the same performance as level 2, At the same time can also clearly say their own name, age and other information; Level 4: The patient is awake, Have the same performance as level 3, It can also accurately identify the surrounding environment, And tell you exactly where you are.
3. In addition to receiving different feeding treatment programs in the PACU, the two groups received the same care and diet program formulated by the same care group.

Record: Patients had fasting serum prealbumin, retinol-binding protein levels, and insulin resistance index on the same day, 1day and 3 days after surgery.

Record: 2 hours, 6 hours and 8 hours postoperative digital scores; bloating, hypoxemia and reflux aspiration occurred 24 hours after surgery.

Record: length of hospitalization, first anal exhaust time, first ambulation time, nausea and vomiting, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective knee replacement surgery.
* The patient gave informed consent.
* Age ≥65 years, Sex is not limited
* American Society of Anesthesiologists (ASA)Ⅰ~Ⅲ level
* Body Mass Index (BMI)18~28kg/m2

Exclusion Criteria:

* Preoperative gastric emptying disorders, such as gastroesophageal reflux or previous surgery.
* Diabetes mellitus, severe renal insufficiency, or other severe metabolic diseases.
* History of motion sickness.
* Mental disorders, alcoholism, or a history of substance abuse.
* Patients with abnormal swallowing function.
* Maltodextrin, fructose allergy or intolerance.
* Surgery time was greater than 3 hours.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Pre-albumin levels at fasting | 1 day after surgery
  The change in prealbumin levels in venous blood in a fasting state in the early morning can reflect whether carbohydrate administration is favorable in the early postoperative period

SECONDARY OUTCOMES:
Pre-albumin levels at fasting | On the day of the surgery
  The change in prealbumin levels in venous blood in a fasting state in the early morning can reflect whether carbohydrate administration is favorable in the early postoperative period
Pre-albumin levels at fasting | 3 days after surgery
  The change in prealbumin levels in venous blood in a fasting state in the early morning can reflect whether carbohydrate administration is favorable in the early postoperative period
Retinol-binding protein levels at fasting levels | Analyzed in early morning fasting venous blood samples at 3 time points： Operatively （day 0）， postoperatively（day1）， postoperatively（day3）
  Changing the levels of early morning retinol-binding protein in venous blood in a fasting state can reflect whether carbohydrate administration is advantageous in the early postoperative period
Insulin resistance index at fasting | Analyzed in early morning fasting venous blood samples at 3 time points： Operatively （day 0）， postoperatively（day1）， postoperatively（day3）
  In the venous blood in an early morning fasting state, the change in the insulin resistance index can reflect whether the carbohydrate administration is favorable in the early postoperative period
The NRS score for the thirst condition | 2 hours, 6 hours and 8 hours after surgery
  Numerical Rating Scale (Numerical Rating Scale, NRS) was used to evaluate patients' thirst, according to a scale of 0 to 10 points: no thirst and 10 points: unbearable thirst. A lower NRS score for thirst conditions indicates that early carbohydrate postoperative administration is advantageous.
The NRS score for the starvation conditions | 2 hours, 6 hours and 8 hours after surgery
  Using the digital scoring method (Numerical Rating Scale, NRS) to assess patient hunger, according to the 0 to 10 scale: no hunger and 10: unbearable hunger. A lower NRS score for starvation conditions indicates that early carbohydrate postoperative administration is advantageous.
The degree of abdominal distension | 24 hours after surgery
  Using grading method, complaining of abdominal distention, tolerable, feeling gas rolling in the abdomen, no obvious abdominal signs, mild abdominal distension, abdominal distention, moderate abdominal distension, vomiting, dyspnea, and significant abdominal bulge.
Time of the first anal exhaust after surgery | Up to 48 hours postoperative
  The advanced time of the first postoperative anal exhaust indicates a favorable early postoperative carbohydrate administration
length of patient stays | Up to 7days postoperative
  The shortened length of hospital stay indicated that early postoperative carbohydrate administration was advantageous
Time of first ambulation after surgery | Up to 48 hours postoperative
  The early time of the first postoperative ambulation indicates that early postoperative carbohydrate administration is advantageous
The incidence of reflux aspiration | 24 hours after surgery
  The reduced incidence of reflux aspiration indicates that early postoperative carbohydrate administration is advantageous
The incidence rate of hypoxemia | 24 hours after surgery
  The reduced incidence of hypoxemia suggests that early postoperative carbohydrate administration is advantageous
Patient satisfaction score | Up to 48 hours postoperative
  Rated on a 0-10 scale, with a higher score representing greater satisfaction.
The incidence and severity of various adverse events (AE) from the start of oral carbohydrates until the end of the trial | Up to 48 hours postoperative
  The lower the incidence and severity of various adverse events (AE) from the start of postoperative oral carbohydrates until the end of the trial, it indicates that the early postoperative carbohydrate administration is beneficial
The incidence and severity of adverse events such as nausea, vomiting and hypoxemia from the first start of drug administration until the end of the trial; | Up to 48 hours postoperative
  The lower the incidence and severity of adverse events such as nausea, vomiting, and hypoxemia until the end of the trial with the initial drug administration indicates that the early postoperative carbohydrate administration is advantageous
Number of antiemetic drugs used within 24h of initial administration until the first start of administration | Up to 24 hours postoperative
  The less use of antiemetic drugs within 24h after the first start of postoperative administration indicates that early postoperative carbohydrate administration is advantageous

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller TE, Roche AM, Mythen M. Fluid management and goal-directed therapy as an adjunct to Enhanced Recovery After Surgery (ERAS). Can J Anaesth. 2015 Feb;62(2):158-68. doi: 10.1007/s12630-014-0266-y. Epub 2014 Nov 13. PMID 25391735
- [Background] Rizvanovic N, Nesek Adam V, Causevic S, Dervisevic S, Delibegovic S. A randomised controlled study of preoperative oral carbohydrate loading versus fasting in patients undergoing colorectal surgery. Int J Colorectal Dis. 2019 Sep;34(9):1551-1561. doi: 10.1007/s00384-019-03349-4. Epub 2019 Jul 15. PMID 31309323
- [Background] Nygren J, Thorell A, Ljungqvist O. Preoperative oral carbohydrate therapy. Curr Opin Anaesthesiol. 2015 Jun;28(3):364-9. doi: 10.1097/ACO.0000000000000192. PMID 25827282
- [Background] [4] Surgery Branch of Chinese Medical Association, Anesthesiology Branch of Chinese Medical Society. Chinese Expert Consensus and Path Management Guidelines for Accelerating Rehabilitation Surgery (2018) [J]. Chinese Journal of Anesthesiology, 2018,38 (001): 8-13.
- [Background] Yang R, Tao W, Chen YY, Zhang BH, Tang JM, Zhong S, Chen XX. Enhanced recovery after surgery programs versus traditional perioperative care in laparoscopic hepatectomy: A meta-analysis. Int J Surg. 2016 Dec;36(Pt A):274-282. doi: 10.1016/j.ijsu.2016.11.017. Epub 2016 Nov 10. PMID 27840308
- [Background] [6] Bethune Orthopaedic Accelerated Rehabilitation Alliance, Bethune Charity Foundation Orthopaedic Professional Committee of trauma, Joint Surgery Professional Committee of Bethune Charity Foundation, etc. Guidelines for the management of perioperative fasting fasting in orthopaedic surgery [J]. Chinese Journal of Trauma and Orthopedics, 2019,21 (10): 829-834.
- [Background] Smith MD, McCall J, Plank L, Herbison GP, Soop M, Nygren J. Preoperative carbohydrate treatment for enhancing recovery after elective surgery. Cochrane Database Syst Rev. 2014 Aug 14;2014(8):CD009161. doi: 10.1002/14651858.CD009161.pub2. PMID 25121931
- [Background] Noba L, Wakefield A. Are carbohydrate drinks more effective than preoperative fasting: A systematic review of randomised controlled trials. J Clin Nurs. 2019 Sep;28(17-18):3096-3116. doi: 10.1111/jocn.14919. Epub 2019 Jun 10. PMID 31112338
- [Background] [9] Wang Cuilan, Huang Yuting, Zeng Qing, et al. Study on postoperative fasting water prohibition time under ERAS concept [J]. Clinical Medical Engineering, 2022,29 (4): 2.

DOCUMENTS (1):
  • Study Protocol (2022-10-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT05603364/Prot_000.pdf